CLINICAL TRIAL: NCT04050176
Title: Use of Blinded Tapering for Hypnotic Discontinuation
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS3239
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Hypnotic Dependence Among Those With Insomnia
Keywords: insomnia; sedative hypnotics; hypnotic tapering
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Two groups: Blinded and Unblinded.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants assigned to Blinded Taper group will not know rate of tapering. Outcomes assessor will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blinded Hypnotic Medication Taper (BT) (Experimental): Participants assigned to the Blinded Taper group will not know the medication dose they receive during the Structured Medication Taper (SMT) phase.
  Interventions: Behavioral: Hypnotic Medication Blinded Taper
- Open-Label Hypnotic Medication Taper (OLT) (Active Comparator): Participants assigned to the Open-Label Hypnotic Medication Taper group will know the medication dose they receive during the SMT phase.
  Interventions: Behavioral: Hypnotic Medication Open-Label Taper

INTERVENTIONS:
Behavioral: Hypnotic Medication Open-Label Taper — Participants will have their soporific hypnotic medication dosage reduced by 25% every two weeks during a 10 week open-label tapering period.
  Other Names: Quarter Drug Open-Label Taper
  Arms: Open-Label Hypnotic Medication Taper (OLT)
Behavioral: Hypnotic Medication Blinded Taper — Participants will have their soporific hypnotic medication dosage reduced by 25% every two weeks during a 10 week blinded tapering period.
  Other Names: Quarter Drug Blinded-Label Taper
  Arms: Blinded Hypnotic Medication Taper (BT)

SUMMARY:
The study will employ a randomized longitudinal clinical trial design to evaluate the relative efficacy of a blinded hypnotic tapering protocol when used in combination with therapist delivered Cognitive Behavioral Therapy for Insomnia (CBTI) for enhancing hypnotic discontinuation rates. A blinded SMT+CBTI intervention will be compared to open-label SMT+CBTI.

DETAILED DESCRIPTION:
Treatment-seeking insomnia sufferers most often present in primary care venues where the first and usually only treatment is a prescription for a sedative hypnotic, typically a benzodiazepine (BZD) or newer benzodiazepine receptor agonist (BzRA). For some patients, short-term or intermittent hypnotic use provides satisfactory insomnia relief. However, more than 65% of individuals who are prescribed hypnotics use them for more than a year, and > 30% remain on these agents for more than five years. Whereas some patients may appreciate partial or full relief of insomnia symptoms with ongoing hypnotic use, continuous long-term use of these agents may not represent optimal therapy. Many insomnia patients who participate in non-drug insomnia therapy such as cognitive behavioral insomnia therapy (CBT-I) achieve sustained insomnia remission long after a time-limited course of treatment. However, it is difficult for most long-term hypnotic users to convert from use of medications to a self-management approach. Interventions that combine CBT-I with supervised medication tapering (SMT) have shown the greatest promise for achieving this outcome, but almost 50% of patients who receive this assistance either fail to discontinue their hypnotics or return to them even if they do achieve short-term abstinence. Our clinical and research observations suggest that psychological factors including sleep-related performance anxiety, low sleep-related self-efficacy and beliefs about needs for medications interact to lead to difficulties abstaining from hypnotic use. Moreover, our highly promising pilot data suggest that such factors may be mitigated by use of a blinded SMT protocol which appears to increase rates of medication abstinence. The current project will use a 2 x 4 randomized longitudinal clinical trial design to test the relative efficacy of our highly promising blinded tapering protocol, vis a vis open-label tapering, when combined with therapist delivered CBT-I. A sample of 260 will be enrolled, complete pre-intervention baseline measures and then be randomly assigned to: (1) a blinded hypnotic SMT + therapist delivered CBT-I; or (2) open-label tapering + CBT-I. During treatment all enrollees will first receive one on one treatment sessions with a trained CBT-I therapist over a 6 week period while maintaining baseline doses of their respective hypnotics. They then will begin a 10 week SMT during which they are provided a blinded or open-label tapering SMT protocol. During this phase they will have their hypnotic medication doses reduced by 25% every two weeks. Immediately after completing the SMT and again at 3- and 6-month follow-ups they will complete study outcome measures. The primary study outcome will be hypnotic discontinuance rates of the two treatment groups. Secondary outcomes include nights of hypnotic use per week, nightly average dosage of hypnotic used in diazepam equivalents as well as scores on sleep quality, daytime fatigue and quality of life. This study will lead to refining guidelines for tapering methods and providing a better understanding of treatment outcome predictors so as to provide more successful, person-centered interventions.

ELIGIBILITY:
Inclusion Criteria:

1. be currently using one or more BZD or newer BzRA hypnotics at bedtime for insomnia management;
2. have been using one or more such agents at least 5 nights/week for at least the past 12 months;
3. express interest in discontinuing hypnotic use and learning to manage their insomnia without medications;
4. report one or more failed attempts to discontinue hypnotic use in the past;
5. provide written consent to participate.
6. have an insomnia severity index score > 10 indicating at least mild insomnia symptoms without sleep medication

Exclusion Criteria:

1. an untreated, or unstable psychiatric disorder as suggested by current active symptoms or a medication regimen that has been changed within the past 2 months;
2. a lifetime diagnosis of any psychotic or bipolar disorder
3. an imminent risk for suicide
4. evidence of alcohol or drug abuse (other than hypnotics) within the past year, since such abuse patterns suggest specialized substance abuse treatment may be indicated
5. unstable or terminal physical illness (e.g., cancer), neurological degenerative disease (e.g., dementia) or sleep disruptive medical condition
6. current use of medications known to cause insomnia (e.g., corticosteroids)
7. screening evidence of circadian rhythm sleep disorder (e.g., delayed sleep phase syndrome) or other sleep disorder (e.g. narcolepsy, idiopathic hypersomnolence, Rapid Eye Movement (REM) behavior disorder) for which CBTI would not represent optimal therapy
8. habitual bedtimes later than 2:00 AM or rising times later than 10:00 AM;
9. consuming > 2 alcoholic beverages/day or any cannabis products at least 5 times/week
10. pregnant women or mothers with care-taking responsibilities for infants due to the sleep-disruption caused by such circumstances
11. clinical or polysomnographic evidence of undiagnosed and untreated restless legs syndrome (RLS), sleep apnea or periodic limb movements (PLMS) that require alternative therapies and would limit participants' responses to CBTI

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Hypnotic Discontinuation Rate As Assessed By Analysis of Study Pharmaceutical Records | 10-week tapering phase
  the proportion of participants in each treatment group who achieve full withdrawal of their BZD/BzRA medication without switching to any alternative prescription medication, used on- (e.g., suvorexant) or off-label (e.g. trazodone) to promote sleep

SECONDARY OUTCOMES:
Nights of Hypnotic use/week | Six-month follow up phase
  Measurement will be taken by analysis of participant reports of the proportion of participants in each tapering group who achieve medication abstinence but subsequently return to hypnotic use by the 6-month follow-up visit
Weekly average dosage of hypnotic used in diazepam equivalents | Six-month follow up phase
  Measurement will be taken by analysis of participant reports of their average weekly medication use within proportion of participants in each tapering group who achieve medication abstinence but subsequently return to hypnotic use by the 6-month follow-up visit.
Use of over the counter sleep aids (e.g. Benadryl) as well as use of substances (alcohol, marijuana) | Six-month follow up phase
  Measurement will be taken by analysis of participant reports of their average weekly medication use within proportion of participants in each tapering group who achieve medication abstinence but subsequently return the use of over the counter sleep aids (e.g. Benadryl) as well as use of substances (alcohol, marijuana) by the 6-month follow-up phase

CONTACTS AND LOCATIONS:
Overall Officials: Jack D Edinger, Ph.D., Principal Investigator — National Jewish Health; Fredrick Wamboldt, M.D., Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data Archives. All data related to the clinical trial will be placed in the public domain in a time frame consistent with NIMH policies. Primary datasets will be made available via CDROM. These datasets will not include any personal identification related to participants or clinical sites beyond the usual numerical keys. Variable dictionaries, detailing variable description, format, value domain and labels, will be produced. Raw data will be exported in comma-separated format, to be readable by all major statistical software. Archives will also include data collection instructions and scoring algorithms for inventories. All reading material will be archived in PDF format.